CLINICAL TRIAL: NCT03184194
Title: A Phase 2 Study of Nivolumab Combined With Daratumumab With or Without Low-dose Cyclophosphamide in Relapsed/Refractory Multiple Myeloma
Brief Title: Nivolumab Combined With Daratumumab With or Without Low-dose Cyclophosphamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Erasmus Medical Center (Other); UMC Utrecht (Other); Maastricht University Medical Center (Other); Meander Medical Center (Other); St. Antonius Hospital (Other); Isala (Other); Albert Schweitzer Hospital (Other); Radboud University Medical Center (Other); University Medical Center Groningen (Other); Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, WCJ van de Donk, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA209-755
Record Dates: First submitted 2017-06-02; First posted 2017-06-12 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Myeloma
Keywords: daratumumab; nivolumab; cyclophosphamide
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab-daratumumab (Experimental): daratumumab 16 mg/kg: 8 times once weekly, then 8 times every 2 weeks; then every 4 weeks; nivolumab: 240 mg every 2 weeks during first 6 cycles, followed by 480 mg every 4 weeks
  Interventions: Drug: nivolumab-daratumumab
- Nivolumab-daratumumab with cylclophosphamide (Experimental): daratumumab 16 mg/kg: weekly for 8 weeks, then Q2W for 16 weeks, ten Q4W thereafter; nivolumab: 240 mg every 2 weeks during first 6 cycles, followed by 480 mg every 4 weeks; low-dose cyclophosphamide 50mg daily on days 1-28 of each 28-day cycle;
  Interventions: Drug: nivolumab-daratumumab with low-dose cyclophosphamide

INTERVENTIONS:
Drug: nivolumab-daratumumab — nivolumab-daratumumab will be given without low-dose cyclophosphamide until progression
  Other Names: Opdivo-darzalex
  Arms: Nivolumab-daratumumab
Drug: nivolumab-daratumumab with low-dose cyclophosphamide — nivolumab-daratumumab with low-dose cyclophosphamide will be given until progression
  Other Names: Opdivo-darzalex with endoxan
  Arms: Nivolumab-daratumumab with cylclophosphamide

SUMMARY:
Evaluation of the effect of nivolumab and daratumumab with or without low-dose cyclophosphamide in patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
Myeloma patients who develop bortezomib and lenalidomide-resistant disease have a very poor survival of only a median of 9 months, indicating that new agents are urgently needed. Recent studies have shown that daratumumab as a single agent is effective and well tolerated in these heavily pretreated MM patients. However, approximately 60% of patients do not achieve a partial response, and ultimately all patients will develop progressive disease during daratumumab therapy. In less pretreated patients daratumumab-based combinations (daratumumab plus lenalidomide-dexamethasone or daratumumab plus bortezomib-dexamethasone) were very effective and well tolerated. Therefore, in this study, the investigators will combine daratumumab with other agents to improve survival of heavily pretreated MM patients.

The PD-1 blocker nivolumab, as single agent, does not induce objective responses but induces stable disease in approximately 67% of relapsed/refractory MM patients. We have recently shown that daratumumab treatment results in increased T cell frequencies by eliminating CD38-positive immune suppressor cells, which probably contributes to the durable responses observed with daratumumab.

Cyclophosphamide, at a dose substantially lower than the maximum tolerated dose, has next to its direct anti-tumor activity serveral other effects including anti-angiogenic effects, induction of changes in the micro-environment, and also improvement of the anti-tumor immune response.

In this study, the investigators will combine two or three immune modulating agents with different mechanisms of action in order to improve the outcome of relapsed/refractory MM patients.

The investigators will evaluate in Part A, nivolumab combined with daratumumab with or without low-dose cyclophosphamide (total 40 patients). Based on efficacy and tolerability, the investigators will treat in Part B 20 additional patients with nivolumab combined with daratumumab either with or without low-dose cyclophosphamide based on tolerability and efficacy data obtained in Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years
2. Subject must have documented multiple myeloma as defined by the criteria below:

   * Monoclonal plasma cells in the bone marrow ≥10% at some point in their disease history or presence of a biopsy proven plasmacytoma.
   * Measurable disease as defined by any of the following:

     * Serum monoclonal paraprotein (M-protein) level ≥5 g/L (0.5 g/dL); or urine M-protein level ≥200 mg/24 hours; or serum immunoglobulin free light chain ≥100 mg/L (10 mg/dL) and abnormal serum immunoglobulin kappa lambda free light chain ratio (See Appendix A)
3. Relapsed or refractory disease. Relapse is defined as progression of disease after an initial response to previous treatment, more than 60 days after cessation of treatment. Refractory disease is defined as <25% reduction in M-protein or progression of disease during treatment or within 60 days after cessation of treatment.
4. Subject had at least 2 prior anti-myeloma regimens. (Note: Induction, bone marrow transplant with or without maintenance therapy is considered one regimen.)
5. Subject has developed lenalidomide-refractory disease during prior treatment with a lenalidomide-containing regimen. Refractory disease is defined as <25% reduction in M-protein or progression of disease during treatment or within 60 days after cessation of treatment.
6. Subject received prior treatment with a proteasome inhibitor-containing regimen for at least 2 consecutive cycles.
7. world health organization (WHO) performance 0, 1, or 2
8. Life expectancy at least 3 months
9. Written informed consent

Exclusion Criteria:

1. Prior therapy with daratumumab or other anti-CD38 therapies
2. Non-secretory myeloma
3. Systemic amyloid light-chain (AL) amyloidosis or plasma cell leukemia (>2.0x109/L circulating plasma cells by standard differential) or Waldenstrom's macroglobulinemia
4. Subject has known meningeal involvement of multiple myeloma
5. Subject has received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before start of treatment. This included subjects who have received a cumulative dose of corticosteroid greater than or equal to the equivalence of 140 mg prednisone or a single dose of corticosteroid greater than or equal to the equivalence of 40 mg/day dexamethasone within the 2-week period before start of treatment.
6. Prior treatment with an anti-PD1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
7. Subject has previously received an allogeneic stem cell transplantation (at any time)
8. Inadequate marrow reserve as defined by a platelet count <75 x 109/L (<50 x 109/L if ≥50% of bone marrow mononucleated cells are plasma cells) or an absolute neutrophil count <1.0 x 109/L
9. a) Subject has known chronic obstructive pulmonary disease (COPD) with an Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.

   b) Subject has known moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification. (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
10. Subject has clinically significant cardiac disease, including:

    * Myocardial infarction within 6 months before Cycle 1, Day 1, or unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV)
    * Cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] Version 4 Grade 2 or higher) or clinically significant ECG abnormalities.
    * Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
11. Significant hepatic dysfunction (total bilirubin >1.5 times normal value (except subjects with Gilbert syndrome, who can have total bilirubin <3.0 mg/dL) or transaminases > 3 times normal value), unless related to myeloma
12. Creatinine clearance <30 ml/min.
13. Known hypersensitivity to components of the investigational products or severe allergic or anaphylactic reactions to humanized products.
14. Subject has any concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, etc.) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
15. Subject is known to be seropositive for human immunodeficiency virus (HIV) or known to have acquired immunodeficiency syndrome (AIDS), or any positive test for hepatitis B or hepatitis C indicating acute or chronic infection.
16. History of active malignancy during the past 3 years, except squamous cell and basal cell carcinomas of the skin and carcinoma in situ of the cervix or breast and incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative, or malignancy that in the opinion of the local investigator, with concurrence with the principal investigator, is considered cured with minimal risk of recurrence within 3 years.
17. Subjects with active interstitial pneumonitis
18. Subjects with active, known or suspected autoimmune disease or inflammatory disorder (including inflammatory bowel disease [eg, colitis, Crohn's disease], systemic lupus erythematosus, Wegener's syndrome, myasthenia gravis, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis, etc.). Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
19. Subjects with a condition (other than MM) requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
20. Subject is known or suspected of not being able to comply with the study protocol (eg, because of alcoholism, drug dependency, or psychological disorder) or the subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments.
21. Pregnant or lactating females
22. Women of childbearing potential not willing to use adequate contraception, defined as hormonal birth control or intrauterine device, during the trial and for 1 year after the last dose of daratumumab or nivolumab or lenalidomide. Men who are sexually active with women of childbearing potential who are not willing to use adequate contraception for the duration of treatment with the study drugs and for 1 year after the last dose of daratumumab or nivolumab or lenalidomide.
23. Peripheral neuropathy of ≥grade 2.
24. History of allergy to study drug components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
overall response rate | active treatment period up to 5 years
  the best response obtained during treatment

SECONDARY OUTCOMES:
incidence of treatment emergent adverse events | active treatment period up to 5 years
  type, frequency and severity of adverse events
progression-free survival | up to 5 years
  time from registration to progression or death from any cause, whichever comes first)
overall survival | up to 5 years
  measured until death from any cause. Patients still alive or lost to follow up are censored at the date they were last known to be alive
tumor expression profile as prognostic factor for response/survival | up to 5 years
  tumor expresssion profile by flow-cytometric detection

CONTACTS AND LOCATIONS:
Overall Officials: Niels van de Donk, MD PhD, Principal Investigator — VUmc
Locations (9):
- Netherlands (9):
  - Rijnstate ziekenhuis, Arnhem, Ge
  - Radboud MC, Nijmegen, Ge
  - MUMC, Maastricht, Li
  - VU University Medical Center, Amsterdam, North Holland
  - UMC Groningen, Groningen, Provincie Groningen
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Meander MC, Amersfoort, Utrecht
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
  - UMC Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Noori S, Verkleij CPM, Zajec M, Langerhorst P, Bosman PWC, de Rijke YB, Zweegman S, VanDuijn M, Luider T, van de Donk NWCJ, Jacobs JFM. Monitoring the M-protein of multiple myeloma patients treated with a combination of monoclonal antibodies: the laboratory solution to eliminate interference. Clin Chem Lab Med. 2021 Aug 16;59(12):1963-1971. doi: 10.1515/cclm-2021-0399. Print 2021 Nov 25. PMID 34392637